CLINICAL TRIAL: NCT01498744
Title: Randomized Controlled Trial of Antibiotics in the Management of Children With Community-Acquired Skin and Soft Tissue Abscess Undergoing Incision and Drainage
Brief Title: Randomized Controlled Trial of Antibiotics in the Management of Children With Community-Acquired Abscess
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was closed due to poor enrollment and lack of interest.
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Katherine Barsness, MD, Attending Physician, Department of Surgery, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB # 2010-14118
Record Dates: First submitted 2011-12-20; First posted 2011-12-23 (Estimated); Results first posted 2016-02-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-01

CONDITIONS: Abscess Soft Tissue; Methicillin-resistant Staphylococcus Aureus (MRSA) Infection; Skin Abscess
Keywords: Skin and Soft Tissue Abscess; Methicillin-resistant Staphylococcus aureus (MRSA); Incision and Drainage; Clindamycin; Trimethoprim-sulfamethoxazole; Skin Infection
MeSH Terms: conditions — Infections; Surgical Wound; Cellulitis | interventions — Clindamycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5 days postoperative antibiotic (Experimental): Based on our preliminary susceptibility data, oral clindamycin (10mg/kg up to 300 mg, every 8 hours) is the first line of antibiotic. Patients allergic or intolerant to clindamycin will receive oral trimethoprim-sulfamethoxazole [bactrim] (5mg/kg trimethoprim up to 160 mg, every 12 hours).
  Interventions: Drug: Oral Clindamycin
- 1 day postoperative antibiotic (Experimental): Based on our preliminary susceptibility data, oral clindamycin (10mg/kg up to 300 mg, every 8 hours) is the first line of antibiotic. Patients allergic or intolerant to clindamycin will receive oral trimethoprim-sulfamethoxazole [bactrim] (5mg/kg trimethoprim up to 160 mg, every 12 hours).
  Interventions: Drug: Oral Clindamycin

INTERVENTIONS:
Drug: Oral Clindamycin — Based on our preliminary susceptibility data, oral clindamycin (10mg/kg up to 300 mg, every 8 hours) is the first line of antibiotic. Patients allergic or intolerant to clindamycin will receive oral trimethoprim-sulfamethoxazole [bactrim] (5mg/kg trimethoprim up to 160 mg, every 12 hours).

SUMMARY:
The purpose of this study is to better understand why children develop methicillin-resistant Staphylococcus aureus (MRSA) skin infections that require surgical drainage and whether antibiotics are helpful after the infection is drained in the operating room.

DETAILED DESCRIPTION:
The emergence of community acquired methicillin-resistant Staphylococcus aureus (MRSA) as a pervasive cause of skin and soft tissue infections has increased the number of children requiring incision and drainage (I&D) procedures and heightened concerns about the optimal treatment strategy. Data on patients with methicillin-sensitive Staphylococcus aureus (MSSA) abscesses, as well as emerging data on children with minor MRSA skin and soft tissue abscesses suggest that I&D alone is sufficient therapy. However, given concerns about the pathogenicity of MRSA infections, many patients who require hospital admission and I&D in the operating room receive postoperative antibiotics. The primary objective of this randomized controlled trial is to compare the effect of 5 days versus 1 day of postoperative antibiotics on the rate of treatment failure following I&D of abscesses in children in the era of pervasive MRSA infection. Secondary outcomes to be measured include incidence of additional skin and soft tissue infections in other body sites and incidence of these infections in family members and household contacts. Prospective data will be collected from wound cultures, as well as from nasal, rectal and skin cultures sent at the time of initial I&D to assess for MRSA carrier status. Finally, survey data will be used to assess epidemiologic risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Children between 1 month and 17 years of age who undergo Incision and Drainage of a skin and soft tissue abscess by a member of the Children's Memorial Hospital pediatric surgery faculty.

Exclusion Criteria:

* Children who developed their infection while hospitalized or within 2 weeks of unrelated hospital discharge will be excluded.
* Children with surgical site infections will be excluded.
* Children with inherent or acquired immunodeficiency, including but not limited to transplant patients and patients on chemotherapy or systemic corticosteroids will be excluded.
* Patients admitted to the Infectious Disease service may be excluded at the discretion of the ID attending.
* Patients who are found to have no discreet fluid collections at the time of attempted incision and drainage will be excluded.
* Patients allergic or intolerant to both bactrim and clindamycin will be excluded.
* Patients with cellulitis greater than 5 cm beyond the lateral margin of the abscess (as determined by intraoperative measurements) will be excluded.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2010-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Barsness, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann and Robert H Lurie Children's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 5 Days Postoperative Antibiotic | 1 Day Postoperative Antibiotic
Started | 22 | 31
Completed | 22 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 Days Postoperative Antibiotic | 1 Day Postoperative Antibiotic | Total
Number analyzed (Participants) | 22 | 31 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 31 | 53
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Gender was not collected before this study was closed | NA — Gender was not collected before this study was closed | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Gender was not collected before this study was closed | NA — Gender was not collected before this study was closed | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  United States | 22 | 31 | 53

OUTCOME MEASURES:

1. Primary Outcome: Clinical Resolution of Skin Abscess at Routine Follow-up Visit 10-14 Days Post Operation.
Time Frame: At office visit 10-14 days post operation
Population: Only participants that had data collected for this outcome measure are included above.
Measure: Number; unit: participants
Arm/Group | 5 Days Postoperative Antibiotic | 1 Day Postoperative Antibiotic
Number analyzed (Participants) | 14 | 19
participants | 0 | 1

2. Secondary Outcome: Additional Skin and Soft Tissue Infections in Patient
Description: The outcome measure was reported by responding to a yes/no
Time Frame: Three timepoints: 10-14 days post operation, 3 months post op, and 9 months post op
Population: Only participants that had data collected for this outcome measure are included here.
Measure: Number; unit: participants
Arm/Group | 5 Days Postoperative Antibiotic | 1 Day Postoperative Antibiotic
Number analyzed (Participants) | 14 | 19
participants
  10-14 Days(n=14,19) | 0 | 2
  90 Day(n=13,15) | 2 | 4
  9 Month(n=10,9) | 2 | 3

3. Secondary Outcome: Additional Skin or Soft Tissue Infections in Household Contacts
Time Frame: Three timepoints: 10-14 days post operation, 3 months post op, and 9 months post op
Population: Only participants that had data collected for this outcome measure are included above.
Measure: Number; unit: participants
Arm/Group | 5 Days Postoperative Antibiotic | 1 Day Postoperative Antibiotic
Number analyzed (Participants) | 13 | 19
participants
  10-14 Days(n=13,19) | 0 | 2
  90 Day(n=13,13) | 2 | 4
  9 Month(n=9,10) | 2 | 2

4. Secondary Outcome: Complication to Antibiotic Regime
Time Frame: Three timepoints: 10-14 days post operation, 3 months post op, and 9 months post op
Population: Only participants that had data collected for this outcome measure are included above.
Measure: Number; unit: participants
Arm/Group | 5 Days Postoperative Antibiotic | 1 Day Postoperative Antibiotic
Number analyzed (Participants) | 14 | 19
participants
  10-14 Days(n=14,19) | 0 | 2
  90 Day(n=0,0) | 0 | 0
  9 Month(n=0,0) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the duration of this study. Study started with IRB approval date of February 23, 2010 and was discontinued (last renewal with IRB expired December 13, 2012)
Arm/Group | 5 Days Postoperative Antibiotic | 1 Day Postoperative Antibiotic
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/31
Other Adverse Events (participants affected / at risk) | 0/22 | 0/31

LIMITATIONS AND CAVEATS:
Inadequate enrollment numbers leading to early termination of study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No